CLINICAL TRIAL: NCT05024422
Title: Lactation Inhibition, the Efficiency of Vitamin B6 Versus Cabergoline- Randomized Controlled Trial
Brief Title: Lactation Inhibition, the Efficiency of Vitamin B6 Versus Cabergoline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0053-21
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Lactation Suppressed
MeSH Terms: interventions — Cabergoline; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of Cabergoline (Active Comparator): one dose of 1mg, up to 24 hours postpartum, or 0.25 mg twice a day for two days
  Interventions: Drug: Cabergoline
- Administration of Vitamin B6 (Active Comparator): 200 mg X 3 per day for a week
  Interventions: Drug: Pyridoxine

INTERVENTIONS:
Drug: Cabergoline — Administration of Cabergoline (one dose of 1mg, up to 24 hours postpartum, or 0.25 mg twice a day for two days)
  Arms: Administration of Cabergoline
Drug: Pyridoxine — Administration of Pyridoxine (200 mg X 3 per day for a week)
  Other Names: Vitamin B6
  Arms: Administration of Vitamin B6

SUMMARY:
Some mothers may seek lactation suppression on personal, social, or medical grounds. To reduce congestion symptoms and shorten the duration of milk production lactation suppression can be done pharmacologic or non-pharmacologic. The most common drug for this purpose is Cabergoline, a dopaminergic agonist, that has significant side effects. Cabergoline is not approved for use in patients with hypertensive disorders, fibrotic diseases, heart problems or liver disease. Vitamin B6 has also been studied for this indication with no significant side effects. All those studies conducted before 1980. There is no current literature on the subject. There are no studies comparing Cabergoline to Vitamin B6 for this indication.

Purpose:

The aim of this study is to test whether Cabergoline is more effective than vitamin B6 for lactation suppression.

method: A prospective randomized study in the maternity ward at Haemek medical center in Afula, Israel.

Postpartum women without contraindication to any one of the treatments, who are interested in a pharmaceutical induced lactation suppression will be divided into two randomized groups:

1. Administration of Cabergoline (one dose of 1mg, up to 24 hours postpartum, or 0.25 mg twice a day for two days)
2. Administration of Vitamin B6 (200 mg X 3 per day for a week)

All women will answer a questionnaire to assess breast congestion, milk leakage and breast pain on days 0, 2, 7 and 14.

ELIGIBILITY:
Inclusion Criteria:

1. Postpartum women who are interested in pharmacologic lactation suppression
2. Women over the age of 18

Exclusion Criteria:

1. Women with known sensitivity to vitamin B6 or Cabergoline
2. Women with hypertensive Disorders or contraindication to Cabergoline.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Lactation suppression | 7 days
reduction of congestion | 14 days
cessation of milk leakage | 14 days
cessation of breast pain | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dayan-Schwartz A, Yefet E, Massalha M, Hosari-Mhameed S, Remer-Gross C, Pasand E, Nachum Z. The efficiency of cabergoline vs pyridoxine for lactation inhibition-a randomized controlled trial. Am J Obstet Gynecol. 2024 May;230(5):561.e1-561.e8. doi: 10.1016/j.ajog.2023.10.009. Epub 2023 Oct 11. PMID 37827268